CLINICAL TRIAL: NCT07201961
Title: Verification of Nellcor™ Pulse Oximetry Device With the Nellcor™ Abbreviated Pulse Oximetry Sensor Line in Adult Volunteers
Brief Title: Nellcor™ Abbreviated Sensor Additional Data Collection
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT25017NQABAD
Record Dates: First submitted 2025-08-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Oxygen Saturation Measurement
Keywords: Hypoxia; Pulse Oximetry; Healthy Volunteer
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: All subjects who meet the inclusion criteria and none of the exclusion criteria will be enrolled into the test group and will participate in data collection with use of the Nellcor™ Pulse Oximetry device with each of the market-released Nellcor™ Pulse Oximetry test sensors.

SUMMARY:
To collect data on a variety of market approved Nellcor™ pulse oximetry sensors with the Nellcor™ Pulse Oximetry device to support the market approval.

DETAILED DESCRIPTION:
The purpose of this study is to collect data on the Nellcor™ Pulse Oximetry device when paired with a variety of Nellcor™ Market Released sensors under invasive, controlled desaturation conditions, to verify Pulse Rate and SpO2 accuracy in a diverse participant population over a specified saturation range.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years of age, and < 51 years of age.
2. Participant is willing and able to comply with study procedures and duration.
3. Participant is willing to sign an ICF.
4. Participant weighs > 40kg (88.2 lb).
5. Participant is a non-smoker or has not smoked within 36 hours prior to the study.
6. Cleared same day health assessment form and health screening
7. Successful perfusion index ulnar/ulnar+radial ratio test (Assessed via the Allen's Test) showing adequate collateral blood flow.

Exclusion Criteria:

1. Participant is considered as being morbidly obese (defined as BMI >39.5).
2. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the sites utilized)
3. Participants of childbearing potential who are pregnant, who are trying to get pregnant, or who have a urine test positive for pregnancy on the day of the study.
4. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
5. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
6. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
7. Participants with known respiratory conditions such as:

   1. uncontrolled / severe asthma
   2. flu or influenza type infection
   3. pneumonia / bronchitis
   4. shortness of breath / respiratory distress
   5. unresolved respiratory or lung surgery
   6. emphysema, COPD, lung disease
   7. recent COVID (last 2 months)
8. Participants with known heart or cardiovascular conditions such as:

   1. Uncontrolled hypertension (systolic pressure >140mmHg, or diastolic pressure >90mmHg on 3 consecutive readings day of screening)
   2. previous cardiovascular surgery
   3. chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
   5. previous heart attack
   6. blocked artery
   7. unexplained shortness of breath
   8. congestive heart failure (CHF)
   9. history of stroke and/or transient ischemic attack
   10. carotid artery disease
   11. myocardial ischemia
   12. myocardial infarction
   13. cardiomyopathy
   14. implantable active medical device such as pacemaker or automatic defibrillator
9. Self-reported health conditions as identified in the Health Assessment Form:

   1. Diabetes
   2. uncontrolled thyroid disease
   3. kidney disease / chronic renal impairment
   4. history of seizures (except childhood febrile seizures)
   5. epilepsy
   6. history of unexplained syncope
   7. recent history of frequent migraine headaches (within the last 2 months)
   8. recent symptomatic head injury (within the last 2 months)
   9. cancer requiring chemotherapy, radiation, or current treatment
   10. participants with known clotting disorders
   11. history of bleeding disorders or personal history of prolonged bleeding from injury
   12. history of blood clots
   13. hemophilia
   14. sickle cell trait or disease
   15. current use of blood thinner: prescription or daily use of aspirin
   16. participants with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
   17. participants with severe allergy to iodine (only applicable if iodine is used)
   18. participants with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
   19. arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site, left or right)
   20. history of clinically significant complications from previous arterial cannulation
   21. unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits
   22. other known health condition, upon disclosure in Health Assessment form
10. Failure of the Allen's Test.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants ≥ 18 and < 51 years of age, with varying skin tones and diversity across ethnicity, race, gender, and sex assigned at birth.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pulse rate accuracy | 2 - 3 hours
  Performance will be determined by calculating the accuracy in terms of root mean square difference (ARMS) comparing the pulse rate measurement from the Nellcor Pulse Oximetry device to the heart rate measurements as obtained by ECG.
Evaluation of saturation accuracy | 2-3 Months
  Performance will be determined by calculating the accuracy in terms of root mean square difference (ARMS) comparing the noninvasive oxygen saturation measurement (SpO2) to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Medtronic Clinical Physiology Lab, Denver, Colorado, United States